CLINICAL TRIAL: NCT05432310
Title: Efficacy and Safety of Cryopreserved Autologous Mobilized Peripheral Blood CD34+ HSPCs Transduced Ex Vivo With the EFS-ADA Lentiviral Vector in Patients With Severe Combined Immune Deficiency Due To Adenosine Deaminase Deficiency
Brief Title: Gene Therapy for Adenosine Deaminase Severe Combined Immune Deficiency Using Peripheral Blood and EFS ADA Vector
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Satiro N De Oliveira, Assistant Professor of Pediatrics, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCLA IRB#21-001814
Record Dates: First submitted 2022-06-04; First posted 2022-06-27 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Adenosine Deaminase Severe Combined Immune Deficiency
Keywords: Gene Therapy; Hematopoietic Stem Cell; Lentiviral Vector; Reduced Intensity Conditioning with Busulfan
MeSH Terms: conditions — Severe combined immunodeficiency due to adenosine deaminase deficiency

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized Phase I/II clinical trial to assess the safety and efficacy of gene therapy for ADA SCID by transplantation of autologous mPB CD34+ hematopoietic stem and progenitor cells (HSPC) transduced by the EFS-ADA lentiviral vector.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous mobilized peripheral blood (mPB) transduced with EFS ADA lentiviral vector (Experimental): Evaluate safety and efficacy of this autologous gene therapy
  Interventions: Combination Product: A cryopreserved formulation of autologous mPB CD34+ hematopoietic stem and progenitor cells transduced ex vivo with the EFS-ADA lentiviral vector encoding the human ADA enzyme

INTERVENTIONS:
Combination Product: A cryopreserved formulation of autologous mPB CD34+ hematopoietic stem and progenitor cells transduced ex vivo with the EFS-ADA lentiviral vector encoding the human ADA enzyme — Autologous transplantation of EFS-ADA lentiviral vector transduced, mPB CD34+ cells by central venous infusion, following reduced intensity conditioning with busulfan

SUMMARY:
The aim of this study is to assess the safety and efficacy of autologous transplantation of hematopoietic stem cells (CD34+ cells) from mobilized peripheral blood (mPB) of ADA-deficient SCID infants and children following human ADA gene transfer by the EFS-ADA lentiviral vector. The level of gene transfer in blood cells and immune function will be measured as endpoints.

DETAILED DESCRIPTION:
The study is open to twenty (20) infants and children diagnosed with ADA-deficient SCID who did not have a medically eligible, human leukocyte antigen (HLA)-identical sibling donor for bone marrow transplantation. The EFS-ADA lentiviral vector with the human ADA complementary DNA (cDNA) will be used to transduce autologous CD34+ cells from Granulocyte Colony Stimulating Factor (G-CSF)/Plerixafor mobilized Peripheral Blood (mPB) of these subjects. The subjects will receive pharmacokinetically-adjusted busulfan reduced intensity conditioning prior to re-infusion of their gene-modified cells. Overall survival at two years is the primary endpoint. During the follow-up phase, the investigators aim to determine whether the cells could engraft and produce mature cells that contain and express the corrected ADA gene in the absence of pegylated adenosine deaminase (PEG-ADA) enzyme replacement therapy (ERT), which will be withheld starting on Day +30 following transplant. Efficacy studies to evaluate the level of immune reconstitution, will be performed in the two years of the study. Patients will be asked to enroll into a long-term follow-up study to reach a total of 15 years follow-up after gene therapy.

ELIGIBILITY:
Inclusion Criteria:

All subjects must fulfill the following criteria to be included in the study:

1. Provision of written informed consent prior to any study related procedures. In this study consent must be provided by the parents/legal guardians and, where applicable according to local laws, a signed assent from the child,
2. Subjects ≥30 days of age,
3. With a diagnosis of ADA-SCID based on:

   Evidence of ADA deficiency, defined as:

   i. Decreased ADA enzymatic activity in erythrocytes, leukocytes, skin fibroblasts, or in cultured fetal cells to levels consistent with ADA-SCID as determined by the reference laboratory, or ii. Identified mutations in ADA alleles consistent with a severe reduction in ADA activity,

   Evidence of ADA-SCID based on either:

   i. Family history of a first order relative with ADA deficiency and clinical and laboratory evidence of severe immunologic deficiency, or ii. Evidence of severe immunologic deficiency in subjects prior to the institution of immune restorative therapy, based on
   1. Lymphopenia (absolute lymphocyte count (ALC) <400 cells/mL) OR absence or low number of T cells (absolute CD3+ count < 300 cells/mL), or
   2. Severely decreased T lymphocyte blastogenic responses to phytohemagglutinin (either <10% of lower limit of normal controls for the diagnostic laboratory, or <10% of the response of the normal control of the day, or stimulation index <10), or
   3. Identification of SCID by neonatal screening revealing low T Cell Receptor Excision Circles (TREC) levels.
4. Ineligible for matched family allogeneic bone marrow (BM) transplantation, defined as the absence of a medically eligible HLA-identical sibling or family donor, with normal immune function, who could serve as an allogeneic bone marrow donor.
5. Females of child-bearing age will be required to provide a negative pregnancy test 30 days prior to Visit 2.
6. Subjects and their parents/legal guardians must be willing and able to comply with study restrictions and to remain at the clinic for the required duration during the study period and willing to return to the clinic for the follow up evaluation as specified in the protocol.

Exclusion Criteria:

Subjects will not be eligible for the study if any of the following criteria is fulfilled:

1. Ineligible for autologous HSCT as per clinical site criteria
2. Other conditions which in the opinion of the Principal Investigator and/or Co Investigators, contraindicate the mobilization of peripheral blood or the leukapheresis process, the administration of busulfan and the infusion of transduced cells, or which indicate an inability of the subject or subject's parent/legal guardian to comply with the protocol
3. Hematologic abnormality, defined as:

   * Anemia (Hb <8.0 g/dl).
   * Neutropenia (ANC <500/mm3). Note: ANC <500 with absence of myelodysplastic syndrome on bone marrow aspirate and biopsy and normal marrow cytogenetics are acceptable for eligibility.
   * Thrombocytopenia (platelet count <50,000/mm3, at any age).
   * Prothrombin time or international normalized ratio (INR) and partial thromboplastin time (PTT) >2 x upper limit of normal (ULN) (subjects with a correctable deficiency controlled on medication will not be excluded).
   * Cytogenetic abnormalities on peripheral blood or bone marrow or amniotic fluid (if available).
   * Prior allogeneic HSCT with cytoreductive conditioning.
4. Pulmonary abnormality, defined as:

   * Resting O2 saturation by pulse oximetry <90% on room air.
   * Chest X-ray indicating active or progressive pulmonary disease. Note: Chest X ray indicating residual signs of treated pneumonitis is acceptable for eligibility.
5. Cardiac abnormality, defined as:

   * Abnormal ECG indicating cardiac pathology.
   * Uncorrected congenital cardiac malformation with clinical symptoms.
   * Active cardiac disease, including clinical evidence of congestive heart failure, cyanosis, hypotension.
   * Poor cardiac function as evidenced by left ventricular ejection fraction <40% on echocardiogram.
6. Neurologic abnormality, defined as:

   * Significant neurologic abnormality revealed by examination.
   * Uncontrolled seizure disorder.
7. Renal abnormality, defined as:

   * Renal insufficiency: serum creatinine ≥1.2 mg/dl (106 µmol/L), or ≥3+ proteinuria.
   * Abnormal serum sodium, potassium, calcium, magnesium or phosphate levels at >2 x ULN.
8. Hepatic/gastrointestinal abnormality, defined as:

   * Serum transaminases >5 x ULN.
   * Serum bilirubin >2 x ULN.
   * Serum glucose >1.5 x ULN.
9. Oncologic disease, defined as:

   * Evidence of active malignant disease other than dermatofibrosarcoma protuberans (DFSP).
   * Evidence of DFSP expected to require anti-neoplastic therapy within the 5 years following the infusion of genetically corrected cells (if anti-neoplastic therapy has been completed, a subject with a history of DFSP can be included).
   * Evidence of DFSP expected to be life limiting within the 5 years following the infusion of genetically corrected cells.
10. Known sensitivity to Busulfan.
11. Confirmation of an infectious disease by deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) positive at time of assessment for the following:

    * HIV-1,
    * Hepatitis B,
    * Parvovirus B19.
12. The subject is pregnant or has a major congenital anomaly.
13. Is likely to require treatment during the study with drugs that are not permitted by the study protocol.
14. The subject has previously received another form of gene therapy.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Survival | 24 months
  The primary study outcome will be to determine survival for all subjects 2 years after gene therapy

SECONDARY OUTCOMES:
Evaluate Safety from clinical adverse events. | 24 months
  Evaluate safety of the treatment by recording clinical adverse events (AE).
Evaluate Safety from replication competent lentivirus by quantitative polymerase chain reaction (qPCR) assay. | 24 months
  Evaluate safety by recording incidents of replication competent lentivirus by qPCR assay..
Evaluate Safety from vector-related clonal expansion by non-restrictive Linear Amplification Polymerase Chain Reaction (nrLAM-PCR) | 24 months
  Evaluate safety by recording incidence of vector-related clonal expansion by nrLAM-PCR
Record event free survival at 24 months | 24 months
  Record Event Free Survival as a definition of "failure" of the therapy. Event-free survival is defined as the proportion of subjects alive with no "event", an "event" being the resumption of PEG-ADA ERT or the need for a rescue allogeneic hematopoietic stem cell transplant (HSCT), or death.
Determine incidence of Infection over two years after gene therapy | 24 months
  Determine the incidence and severity of infections post-gene therapy (subsequent to hematopoietic reconstitution). Over 2 years, record the incidence of hospitalizations or outpatient-based treatments for systemic bacterial, fungal, or viral infections (including, but not limited to Cytomegalovirus (CMV) infections).
Neuro-developmental Outcomes by neurodevelopmental testing (subjects 5-7 yeas of age) | 24 months
  Measure neuro-developmental status post-gene therapy. Perform age-appropriate neuro-developmental assessments testing (5- 7 years of age) at baseline and 2 years post-gene therapy - Wechsler Scale of Intelligence
Neuro-developmental Outcomes by neurodevelopmental testing (subjects 1 year -42 month of age) | 24 months
  Measure neuro-developmental status post-gene therapy. Perform age-appropriate neuro-developmental assessments testing (1 year to 42 months of age) at baseline and 2 years post-gene therapy - : Bayley Scale of Infant Development
Neuro-developmental Outcomes by Brain Stem Evoked Response (BAER) testing | 24 months
  Measure neuro-developmental status post-gene therapy - Perform Brainstem Auditory Evoked Response test at baseline and at 2 years.
Cessation of immunoglobulin replacement therapy (IgRT). | 24 months
  Record time post-gene therapy that immunoglobulin replacement therapy (IgRT) is stopped based on defined criteria.

OTHER OUTCOMES:
Exploratory Study Objectives to measure biological correlates of efficacy - Vector Copy Number (VCN) in peripheral blood leukocytes | 24 months
  The Exploratory Study Objectives are to measure biological correlates of efficacy.
  1. Quantify gene marking by vector copy number (VCN) in peripheral blood leukocytes by droplet digital polymerase chain reaction (ddPCR).
Exploratory Study Objectives to measure biological correlates of efficacy (Vector integrant diversity) | 24 months
  The Exploratory Study Objectives are to measure biological correlates of efficacy.
  2. Quantify clonal diversity of vector integrants by non-restrictive Linear Amplification polymerase chain reaction (nrLAM-PCR). nrLAM-PCR identifies all distinct vector integrants in a cell sample from patients. The presence of >1,000 unique integration sites in a sample indicates diversity of hematopoietic stem cell of clonal engraftment
Exploratory Study Objectives to measure biological correlates of efficacy (expressed ADA enzyme in erythrocytes) | 24 months
  The Exploratory Study Objectives are to measure biological correlates of efficacy.
  3. Measure ADA enzyme activity in erythrocytes as an indicator of expression of functional ADA enzyme from the vector.
Exploratory Study Objectives to measure biological correlates of efficacy Deoxyadenosine nucleotides in erythrocytes) | 24 months
  The Exploratory Study Objectives are to measure biological correlates of efficacy.
  4. Measure total deoxyadenosine nucleotides in erythrocytes.
Exploratory Study Objectives to measure biological correlates of efficacy (Immune reconstitution - quantify T and B cell) | 24 months
  The Exploratory Study Objectives are to measure biological correlates of efficacy.
  5. Assess immune reconstitution by measuring absolute numbers of T and B cells .
Exploratory Study Objectives to measure biological correlates of efficacy (Immune reconstitution - measure serum immunoglobulins) | 24 months
  The Exploratory Study Objectives are to measure biological correlates of efficacy.
  6. Assess immune reconstitution by measuring serum immunoglobulin levels
Exploratory Study Objectives to measure biological correlates of efficacy (Immune reconstitution - response to tetanus vaccine) | 24 months
  The Exploratory Study Objectives are to measure biological correlates of efficacy.
  7. Assess immune reconstitution by measuring response to tetanus vaccine by measuring serum anti-tetanus antibody titers after tetanus vaccination
Exploratory Study Objectives to measure biological correlates of efficacy Parent report Quality of Life | 24 months
  The Exploratory Study Objectives are to measure biological correlates of efficacy.
  8. Parent-Reported Quality of Life (PedsQL 4.0) at baseline and 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Satiro De Oliveira, MD, Principal Investigator — Assistant Professor
Locations (1):
- University of California, Los Angeles (UCLA), Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kohn DB, Booth C, Shaw KL, Xu-Bayford J, Garabedian E, Trevisan V, Carbonaro-Sarracino DA, Soni K, Terrazas D, Snell K, Ikeda A, Leon-Rico D, Moore TB, Buckland KF, Shah AJ, Gilmour KC, De Oliveira S, Rivat C, Crooks GM, Izotova N, Tse J, Adams S, Shupien S, Ricketts H, Davila A, Uzowuru C, Icreverzi A, Barman P, Campo Fernandez B, Hollis RP, Coronel M, Yu A, Chun KM, Casas CE, Zhang R, Arduini S, Lynn F, Kudari M, Spezzi A, Zahn M, Heimke R, Labik I, Parrott R, Buckley RH, Reeves L, Cornetta K, Sokolic R, Hershfield M, Schmidt M, Candotti F, Malech HL, Thrasher AJ, Gaspar HB. Autologous Ex Vivo Lentiviral Gene Therapy for Adenosine Deaminase Deficiency. N Engl J Med. 2021 May 27;384(21):2002-2013. doi: 10.1056/NEJMoa2027675. Epub 2021 May 11. PMID 33974366
- [Background] Carbonaro DA, Zhang L, Jin X, Montiel-Equihua C, Geiger S, Carmo M, Cooper A, Fairbanks L, Kaufman ML, Sebire NJ, Hollis RP, Blundell MP, Senadheera S, Fu PY, Sahaghian A, Chan RY, Wang X, Cornetta K, Thrasher AJ, Kohn DB, Gaspar HB. Preclinical demonstration of lentiviral vector-mediated correction of immunological and metabolic abnormalities in models of adenosine deaminase deficiency. Mol Ther. 2014 Mar;22(3):607-622. doi: 10.1038/mt.2013.265. Epub 2013 Nov 20. PMID 24256635